CLINICAL TRIAL: NCT04916028
Title: Clinical Characteristics of Patients Referred to a Substance Abuse Liaison Department in an Academic Hospital, France
Acronym: AddictUrge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0092
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Substance Abuse; Emergencies; Personality Disorders; Substance Use Disorders
Keywords: Substance abuse liaison-department; Emergencies; Academic Hospital; Personality Disorders; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders; Emergencies; Personality Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Coalition on Psychiatric Emergencies (CPE) stressed in 2016 that emergency providers were increasingly recognizing the important role of the Emergency Department (ED) in reducing adverse outcomes associated with untreated with substance abuse liaison department (SUDs). Additional research is required to close identified knowledge gaps and improve care of ED patients with SUD. Of the more than 4.5 million ED visits in 2009 in US for drug-related causes,34-32% involved alcohol use alone or in combination with other drugs. Few studies investigated the clinical characteristics of patients referred to an addiction liaison department in a general hospital. The present study will be retrospective in a sample of 700 patients consecutively admitted for addictive behaviors in the emergency department and in the Medicine or Surgery departments of the Amiens University Hospital Center, France.

ELIGIBILITY:
Inclusion Criteria:

* patient addressed to University Hospital Emergency Department and consecutively referred to a substance abuse liaison department in the Amiens Academic Hospital, France between 2017 and 2020.
* Patients must be able to speak French

Exclusion Criteria:

* Neurological disorders
* patients who are not able to speak French

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients consecutively admitted for addictive behaviors in the emergency department and in the Medicine or Surgery departments of the Amiens University Hospital Center, France.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
sociodemographic characteristics of patients referred to an addiction liaison department in a Academic general hospital | one month
clinical characteristics of patients referred to an addiction liaison department in a Academic general hospital | one month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No